CLINICAL TRIAL: NCT01403194
Title: Impact of Treatment of Sleep Disordered Breathing With Continuous Positive Airway Pressure (CPAP) on Cardiometabolic Risk Markers
Brief Title: Continuous Positive Airway Pressure and Cardiometabolic Risk
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Analysis was not done because only 1 subject was able to come back for the 3 month follow up visit.
Sponsor: Mayo Clinic (Other)
Responsible Party: Seema Kumar, MD, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 10-004698
Record Dates: First submitted 2011-04-06; First posted 2011-07-27 (Estimated); Results first posted 2014-05-13 (Estimated); Last update posted 2014-05-13 (Estimated); Status verified 2014-04

CONDITIONS: Sleep Disordered Breathing
Keywords: Sleep Disordered Breathing; CPAP; BiPAP; Cardiovascular risk markers
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CPAP/Bi-PAP (Experimental): Subjects will be treated with either CPAP or Bi-PAP for three months.
  Interventions: Device: CPAP/BiPAP

INTERVENTIONS:
Device: CPAP/BiPAP — Subjects will be treated with either CPAP or Bi-PAP for three months.

SUMMARY:
The hypothesis for this study is that children with sleep disordered breathing will benefit from treatment with Continuous Positive Airway Pressure (CPAP) or Bi-level Positive Airway Pressure (BiPAP) in terms of reduction in cardiovascular risk markers and insulin resistance.

The CPAP machine delivers a predetermined level of pressure. It releases a stream of compressed air through a hose to the nose mask and keeps the upper airway open under continuous air pressure. This air pressure prevents obstructive sleep apnea, which occurs as a result of narrowing of the airway due to the relaxation of upper respiratory tract muscles during sleep. This machine helps to increase the oxygen flow by keeping the airway open.

The BiPAP machine delivers two levels of pressure. Inspiratory Positive Airway Pressure (IPAP) is a high amount of pressure, applied when the patient inhales and a low Expiratory Positive Airway Pressure (EPAP) during exhalation.

DETAILED DESCRIPTION:
Obese children with Moderate to Severe Sleep Apnea will have baseline evaluation of markers of cardiometabolic risk and insulin resistance. Subjects will then use either the CPAP or BiPAP machine for 3 months and will return for another blood draw for measurement of the markers for cardiometabolic risk and insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

1. Body mass index greater than 95th percentile for age and gender
2. Moderate to severe obstructive sleep apnea (OSA) (as defined by an apnea-hypopnea index (AHI) score of ≥5 events per hour).

Only patients who provide informed assent or consent and also have consent from a parent will be included.

Exclusion Criteria:

1. Predominant central sleep apnea
2. Type 1 Diabetes
3. Type 2 Diabetes
4. Requires use of supplemental oxygen
5. Active infection, cancer, or chronic inflammatory disorder
6. Use of systemic steroids
7. Simultaneous use of peroxisome proliferator-activated receptor (PPAR)-alpha (e.g., gemfibrozil, fenofibrate) or PPAR-gamma (e.g., rosiglitazone, pioglitazone)

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 11 (Actual)
Dates: Start 2011-03; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Seema Kumar, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 11 subjects with a high probability of Obstructive Sleep Apnea (OSA) were consented, and all had a baseline blood draw. 2 subjects had a normal sleep study. 9 subjects had a polysomnogram suggestive of OSA, and were given the intervention of 3 months of Continuous Positive Airway Pressure (CPAP) or Bi-Level Positive Airway Pressure (Bi-PAP) use.
Period: Overall Study
Arm/Group | CPAP/Bi-PAP
Started | 11
Completed | 1
Not Completed | 10
Not completed — Screen Failure | 2
Not completed — Lost to Follow-up | 8

BASELINE CHARACTERISTICS:
Arm/Group | CPAP/Bi-PAP
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Change in Level of Fasting Glucose
Time Frame: baseline, 3 months
Population: Only one participant returned for the 3 month visit.
Arm/Group | CPAP/Bi-PAP
Number analyzed (Participants) | 0

2. Secondary Outcome: Change in Level of Fasting Insulin
Time Frame: baseline, 3 months
Population: Only one participant returned for the 3 month visit.
Arm/Group | CPAP/Bi-PAP
Number analyzed (Participants) | 0

3. Secondary Outcome: Change in Level of Lipids
Time Frame: baseline, 3 months
Population: Only one participant returned for the 3 month visit.
Arm/Group | CPAP/Bi-PAP
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | CPAP/Bi-PAP
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

LIMITATIONS AND CAVEATS:
Analysis was not done because only 1 subject was able to come back for the 3 month follow up visit.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No